CLINICAL TRIAL: NCT01851057
Title: Supporting Treatment Adherence Regimens in Pediatric Epilepsy: The STAR Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD073115 (NIH); R01HD073115 (NIH)
Record Dates: First submitted 2013-05-01; First posted 2013-05-10 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2019-01

CONDITIONS: Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education Only (Active Comparator): Education only arm (8 total sessions)
  Interventions: Behavioral: Education Only
- STAR: Education and Problem Solving (Experimental): Problem-solving and education intervention (8 total sessions)
  Interventions: Behavioral: STAR

INTERVENTIONS:
Behavioral: STAR — Problem-solving and education intervention (8 total sessions)
  Arms: STAR: Education and Problem Solving
Behavioral: Education Only — Education around epilepsy (8 total sessions)
  Arms: Education Only

SUMMARY:
Fifty-eight percent of children with new-onset epilepsy do not take their antiepileptic drugs (AEDs) as prescribed (i.e., non-adherence). Non-adherence, which is modifiable, is associated with continued seizures, mortality, poor quality of life, and high healthcare costs. There are no adherence interventions for young children with epilepsy and their families; thus, the current proposal examines a family-based behavioral treatment focused on improving epilepsy knowledge and problem-solving around barriers to adherence in young children with epilepsy and their families with the goal of improving adherence and ultimately, seizures and quality of life. It is hypothesized that children with newly diagnosed epilepsy and their families who participate in the problem-solving intervention will have significant improvements on adherence compared to those in the education only intervention.

DETAILED DESCRIPTION:
Non-adherence to antiepileptic drugs (AEDs) is a common (i.e., 58% of patients have some level of non-adherence) and previously under-recognized problem for young children with newly diagnosed epilepsy. This is surprising given the consequences of non-adherence in patients with epilepsy are extremely serious, including continued seizures, mortality, and high healthcare expenditures. Despite the critical need to develop and implement interventions to improve adherence, there are no family-based interventions for young children with epilepsy and their families. As such, we developed a family-tailored adherence intervention (STAR: Supporting Treatment Adherence Regimens) focused on increasing epilepsy knowledge and problem-solving skills around barriers to adherence for children with epilepsy and their families. Data from our pilot adherence intervention studies demonstrated good preliminary effects (effect size= 0.64) and excellent feasibility, with families reporting that the intervention was beneficial and a positive experience for their family. Capitalizing on these findings, the next logical step is to test the efficacy of the STAR intervention to improve AED adherence in 200 children with epilepsy via a randomized controlled trial. Thus, the aims of the study are to examine the short-term and long-term effects of the STAR intervention on electronically-monitored medication adherence in children with new-onset epilepsy compared to an education only (EO) intervention. In addition, exploratory aims are to examine the effect of the STAR intervention on seizure freedom and QOL in children with epilepsy compared to the EO intervention. The current study uses an innovative, sequential, randomization enrichment design that preventatively targets 200 patients with new-onset epilepsy, between 2-12 years, who demonstrate non-adherence. Using criteria established from our pilot studies, adherence falling below 95% within the first six months of the study will trigger participant randomization into one of two 8-session interventions: STAR or EO. If the aims of the project are achieved, this study will change the practice of pediatric epilepsy by providing a proven approach to the routine monitoring and treatment of AED non-adherence in epilepsy clinics across the nation. This study also lays the foundation for determining the long term impact of adherence intervention on morbidity and mortality. In addition, this study's innovative methodological enrichment design should be generalizable to other pediatric conditions and lead to the development of cost effective, clinic-based adherence promotion interventions.

ELIGIBILITY:
Inclusion Criteria:

* ages 2-12 years
* diagnosis of epilepsy within approximately 6 months
* only one prescribed AED
* family lives < 75 miles from Cincinnati Children's Hospital Medical Center (CCHMC)
* ability to read English

Exclusion Criteria:

* comorbid medical disorders requiring daily medication
* parent-reported significant developmental delays (e.g. Autism)
* liquid AED formulation due to electronic monitoring incompatibility.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Adherence rate (short-term) | 30 day post intervention adherence rate
  This is a measure of adherence, using an electronic monitor called the Medication Event Monitoring System (MEMS) TrackCap, and adherence rates range from 0 to 100%. Adherence rates will be calculated at baseline and represent a rate from 0 to 100. Similarly, an adherence rate will be calculated for the 30 day post intervention period, with a rate between 0-100%. The change score for the mean of the 30 days of adherence immediately following the end of intervention relative to the mean adherence obtained during the30 day screening period will be calculated.

SECONDARY OUTCOMES:
Adherence rate (long-term) | 3, 6 and 12 months post intervention
  This is a measure of adherence, using an electronic monitor called the MEMS TrackCap, and adherence rates range from 0 to 100%. The outcome will be a comparison of baseline 30 day adherence, which ranges from 0 to 100%, to the 3, 6, and 12 month post intervention adherence to antiepileptic drugs (0-100%). A change score will be calculated between the baseline and long-term end points of 3, 6 and 12 months.

OTHER OUTCOMES:
Health related quality of life | 6 and 12 months post intervention
  Compare baseline quality of life scores (0-100), based on the PedsQL (Pediatric Quality of Life) questionnaire, compared to 6 and 12 months post intervention.
Seizure absence/presence | 6 and 12 months post intervention
  Compare seizure absence/presence (0=no;1=yes) from baseline to 6 and 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Avani C Modi, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Not being shared

REFERENCES:
- [Derived] Williford DN, Guilfoyle SM, Modi AC. Demystifying a family-based epilepsy adherence problem-solving intervention: Exploring adherence barriers and solutions. Clin Pract Pediatr Psychol. 2023 Mar;11(1):66-73. doi: 10.1037/cpp0000436. Epub 2022 Feb 3. PMID 36969546
- [Derived] Al-Aqeel S, Gershuni O, Al-Sabhan J, Hiligsmann M. Strategies for improving adherence to antiepileptic drug treatment in people with epilepsy. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD008312. doi: 10.1002/14651858.CD008312.pub4. PMID 33089492